CLINICAL TRIAL: NCT05294965
Title: Beta 2 Adrenergic Stimulation vs Cold Exposure to Activate Human Brown Adipose Tissue
Acronym: ASCENT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EKNZ 2022-00037
Record Dates: First submitted 2022-02-09; First posted 2022-03-24 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Thermogenesis
Keywords: brown adipose tissue; beta2-adrenergic agonist; cold exposure
MeSH Terms: interventions — Fenoterol

STUDY DESIGN:
Intervention Model Description: Open-label, cross-over trial in healthy volunteers with random sequence of the two study interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal weight (Experimental): 1. A bolus of 25µg fenoterol will be slowly injected intravenously during 2-3 minutes followed by a continuous infusion of fenoterol 1µg/min over 120 minutes. The total dose of fenoterol per subject will thus be 145µg.
  2. Mild cold exposure: During 120 minutes the water temperature in cooling sleeves, covering the participant's waist, is gradually decreased to 10 degrees or to the lowest tolerable temperature without shivering.
  Interventions: Drug: Fenoterol; Other: Mild cold exposure
- Overweight (Experimental): 1. A bolus of 25µg fenoterol will be slowly injected intravenously during 2-3 minutes followed by a continuous infusion of fenoterol 1µg/min over 120 minutes. The total dose of fenoterol per subject will thus be 145µg.
  2. Mild cold exposure: During 120 minutes the water temperature in cooling sleeves, covering the participant's waist, is gradually decreased to 10 degrees or to the lowest tolerable temperature without shivering.
  Interventions: Drug: Fenoterol; Other: Mild cold exposure

INTERVENTIONS:
Drug: Fenoterol — Intravenous infusion
  Other Names: beta2 adrenoreceptor agonist
Other: Mild cold exposure — Body surface cooling

SUMMARY:
The purpose of the study is to asses brown adipose tissue activity in humans after intravenous administration of the selective beta-2-adrenergic agonist fenoterol as compared to the natural activator of brown adipose tissue, a mild cold stimulus.

DETAILED DESCRIPTION:
The activation of brown adipose tissue in response to beta-2-adrenergic stimulation as compared to cold exposure will be studied in an open-label, cross-over trial in healthy volunteers with random sequence of the two study interventions a) and b):

1. A bolus of 25µg fenoterol will be slowly injected intravenously during 2-3 minutes followed by a continuous infusion of fenoterol 1µg/min over 120 minutes. The total dose of fenoterol per subject will thus be 145µg.
2. During 120 minutes participants will be exposed to a mild cold stimulus water using cooling sleeves, covering the participant's waist, is gradually decrease body surface temperature to 10 degrees or to the lowest tolerable temperature without shivering.

Energy expenditure will be measured during both interventions by indirect calorimetry and brown adipose tissue activity will determined by 18F-FDG-PET/CT 30 min after injection of 75 MBq of 18F-FDG.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18,5-23 kg/m2 or 30-35 kg/m2

Exclusion Criteria:

* History or signs of any medical or psychological condition
* pregnancy or lactation
* medications except prescription free analgesics and contraceptives
* habitual alcohol or tobacco use
* weight change >5% within prior 3 months
* Resting heart rate >85 bpm
* Systolic blood pressure >140 mmHg or diastolic blood pressure <50 mmHg
* Presence of following ECG changes: ST-segment deviations, QTc >500ms, signs of pre-excitation
* Hyper- or Hypothyroidism
* inability to follow study procedures
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* hypersensitivity to cold
* enrolment into study with ionizing radiation within prior 12 months.
* Cold induced thermogenesis of less than 5% basal metabolic rate and normal weight or cold induced thermogenesis of more than 5% and overweight (determined during screening visit)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
BAT SUVmean | 30 minutes after end of intervention
  18F-FDG uptake into the supra-clavicular brown adipose tissue as determined by 18F-FDG PET-CT after the respective study intervention

SECONDARY OUTCOMES:
BAT SUVmax | 30 minutes after intervention
  maximum SUV in supraclavicular adipose tissue (according to BARCIST 1.0)
BAT Volume | 30 minutes after intervention
  volume of supraclavicular adipose tissue (according to BARCIST 1.0)
BAT glycolytic volume | 30 minutes after intervention
  volume of supraclavicular adipose tissue x SUVmean (according to BARCIST 1.0)
Change in energy expenditure | First and last 30 minutes of intervention
  Quantitative change in EE above resting metabolic rate in response to the respective study intervention. Measured by indirect calorimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Betz, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Dept. of Endocrinology, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No